CLINICAL TRIAL: NCT01297855
Title: Randomized Controlled Trial of Colistin Versus Colistin Plus Rifampicin in MDR P.Aeruginosa and A.Baumanii
Brief Title: Colistin Plus Rifampicin in MDR P. Aeruginosa and A. Baumanii
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Visanu Thamlikitkul, Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkok, Thailand, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SirirajCEU51-001
Record Dates: First submitted 2009-07-20; First posted 2011-02-17 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Drug Safety
MeSH Terms: interventions — Colistin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colistin (Active Comparator): Colistate
  Interventions: Drug: Colistin
- Colistin plus Rifampicin (Experimental): Colistate Rifampin
  Interventions: Drug: Colistin plus Rifampicin

INTERVENTIONS:
Drug: Colistin — Colistimethate Sodium dose 2.5-5mg/kg/day
  Other Names: Colistate
  Arms: Colistin
Drug: Colistin plus Rifampicin — Colistin 2.5 to 5 mg/ Kg/ day Rifampin 10 mg/ Kg/ day
  Other Names: Colistate; Rifampin
  Arms: Colistin plus Rifampicin

SUMMARY:
In Siriraj Hospital, Colistin alone for treatment of MDR. A.baumanii or P.aeruginosa contributed to mortality 45%. In vitro studies revealed synergism of Rifampicin and Colistin.

In this study, patients with documented MDR. P.aeruginosa or A.baumanii will be allocated to receive Colistin alone and another group will receive Colistin plus Rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Hospitalized to Siriraj Hospital
* Infection with MDR A.baumanii or P.aeruginosa
* Nescessary for treatment with Colistin
* Patient agrees to participate by giving written informed consent.

Exclusion Criteria:

* pregnancy or lactating mother
* Colistin or Rifampicin allergy
* Active hepatic disease or abnormal liver function test
* patient who suspected infection with mycobacterium tuberculosis
* patient who can not drug by enteral feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
number of subjects with cure or improvement | up to day 28
  Cure Improvement Worse Death

SECONDARY OUTCOMES:
number of subjects with eradication of causative bacteria | up to day 28
  Eradication Persistence Superinfection

CONTACTS AND LOCATIONS:
Overall Officials: Sukij Piyasirisilp, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Infectious disease and Tropical Medicine, Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand